CLINICAL TRIAL: NCT07306377
Title: Helicobacter Pylori Infection as A Potential Risk Factor for Dyslipidemia: Insights From Atherogenic Index of Plasma (AIP)
Brief Title: H. Pylori Infection and AIP Levels
Acronym: HP-AIP
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Nahla Ahmed Khalaf, Lecturer of Tropical Medicine and Infectious Diseases, Tanta University
Other Study IDs: Helicobacter Pylori and AIP
Record Dates: First submitted 2025-12-12; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: H Pylori Infection; Atherogenic Plasma Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1A: H. pylori Positive - Normal AIP Group 1B: H. pylori Positive - Elevated AIP Group 2: H.
  Interventions: Diagnostic Test: urea breath test
- Group 1A: H. pylori Positive - Normal AIP, 1B: H. pylori Positive - Elevated AIP, Group 2: H.
  Interventions: Diagnostic Test: urea breath test

INTERVENTIONS:
Diagnostic Test: urea breath test — Participants will undergo a urea breath test to confirm H. pylori infection status.
  Fasting blood samples will be collected to measure triglycerides and HDL cholesterol, and the Atherogenic Index of Plasma (AIP) will be calculated.

SUMMARY:
Helicobacter pylori is a common bacterial infection of the stomach that can cause ulcers and other digestive problems. Recent studies suggest that this infection may also affect metabolism and blood fats (lipids), which are important for heart health. Changes in lipid levels, such as higher triglycerides and lower "good" cholesterol (HDL), can increase the risk of cardiovascular disease.

This study will examine whether H. pylori infection is linked to changes in lipid profiles, especially the Atherogenic Index of Plasma (AIP). AIP is a calculation based on triglycerides and HDL cholesterol that helps predict the risk of heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Able to sign the written consent.
* Willing to participate in the research and undergo H. pylori testing. Exclusion criteria
* Unwilling to participate in the study.
* History of severe metabolic disorders.
* Taking medications that affect adipose tissue metabolism.
* History of gastric surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) attending the Gastroenterology Unit at Tanta University Hospitals (Egypt) and the Internal Medicine Department at Tadawi Hospital (Saudi Arabia). Participants will include both men and women diagnosed with or without H. pylori infection, recruited consecutively during routine clinical visits.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Atherogenic Index of Plasma (AIP) | Baseline (single fasting blood sample at enrollment).
  AIP is calculated as log10(triglycerides/HDL cholesterol).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided